CLINICAL TRIAL: NCT03035032
Title: A Phase IV Interventional Safety Study of ELIGARD® in Prostate Cancer Patients in Asia (ELIGANT)
Brief Title: A Study of ELIGARD® in Hormone-dependent Prostate Cancer Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Singapore Pte. Ltd. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7015-MA-3072
Record Dates: First submitted 2017-01-25; First posted 2017-01-27 (Estimated); Results first posted 2020-12-09 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-10

CONDITIONS: Prostate Cancer
Keywords: Leuprolide acetate; Prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Leuprolide; luprolide acetate gel depot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Leuprolide Acetate 22.5 milligrams (mg) (Experimental): Participants received 22.5 mg of leuprolide acetate (eligard) by subcutaneous injection at baseline, month 3, 6, 9, 12 and 15.
  Interventions: Drug: Leuprolide

INTERVENTIONS:
Drug: Leuprolide — Subcutaneous Injection
  Other Names: Eligard

SUMMARY:
The objective of this study was to evaluate the safety profile of ELIGARD® in ethnic Asian prostate cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* A patient for whom the physician has decided to initiate treatment with a Luteinizing Hormone Releasing Hormone (LHRH) agonist in standard clinical practice
* Biopsy-proven prostate adenocarcinoma
* Locally advanced prostate cancer with biochemical relapse radical prostatectomy and/or radiotherapy, OR hormonal treatment-naive advanced or metastatic prostate cancer patient who has not received chemotherapy and has no plans to undergo treatment with chemotherapy at study entry.
* Patient who indicates that once the study is completed, he expects having access to androgen deprivation therapy (ADT), either medical or surgical, within the local healthcare system (either through public/ private health insurance or out of pocket payment).

Exclusion Criteria:

* Patient with castrate resistant prostate cancer
* Patient who previously underwent bilateral orchiectomy
* Patient who has received prior treatment with LHRH analogues
* Prior or concomitant treatment with systemic chemotherapy. A patient where there is a likelihood to receive systemic chemotherapy should not be enrolled
* Life expectancy of < 1 year due to comorbidities
* Participation in another interventional clinical trial within one month prior to study entry or during the duration of the study
* Patient who plans to receive intermittent ADT at the time of study entry
* Patient receiving non-palliative radiotherapy within 3 months prior to study entry
* Patient receiving adjuvant ADT in combination with definitive radiotherapy
* Patient with metastatic hormonal treatment-naive prostate cancer, for whom chemo-hormonal treatment (combination of Docetaxel and ADT) is indicated.
* Patient with hypersensitivity to gonadotropin releasing hormone (GnRH), GnRH agonist analogs or any of the components of ELIGARD®
* Patient with any contraindication for ELIGARD® use based on local prescribing information

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2017-06-23 (Actual); Primary Completion 2019-11-19 (Actual); Study Completion 2019-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (19):
- Hong Kong (2):
  - Site HK01001, Hong Kong
  - Site HK01002, Hong Kong
- Site ID02001, Jakarta, DKI Jakarta, Indonesia
- Malaysia (2):
  - Site MY03002, Batu Caves, Selangor
  - Site MY03001, Kuala Lumpur
- Philippines (3):
  - Site PH04001, Makati City, National Capital Region
  - Site PH04003, Manila, National Capital Region
  - Site PH04002, San Juan City, National Capital Region
- Singapore (3):
  - Site SG05001, Singapore
  - Site SG05002, Singapore
  - Site SG05003, Singapore
- Taiwan (3):
  - Site TW06001, Taichung
  - Site TW06002, Taichung
  - Site TW06003, Taipei
- Thailand (3):
  - Site TH07004, Hat Yai, Changwat Songkhla
  - Site TH07001, Muang, Chiang Mai
  - Site TH07003, Bangkok
- Vietnam (2):
  - Site VN08001, Ho Chi Minh City
  - Site VN08002, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Malek R, Wu ST, Serrano D, Tho T, Umbas R, Teoh J, Lojanapiwat B, Ong TA, On WK, Thai SM, Kim J, Pophale R, Chiong E. ELIGANT: a Phase 4, interventional, safety study of leuprorelin acetate (ELIGARD(R)) in Asian men with prostate cancer. Transl Androl Urol. 2022 Feb;11(2):179-189. doi: 10.21037/tau-21-723. PMID 35280654
- See also: Link to results on the Astellas Clinical Study Results website. — https://astellasclinicalstudyresults.com/hcp/study.aspx?ID=395

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Asian male participants above the age of 18 years with biopsy-proven prostate adenocarcinoma who fulfill the eligibility criteria were enrolled in this study.
Pre-assignment Details: 107 participants were enrolled and 106 participants received treatment.
Period: Overall Study
Arm/Group | Leuprolide Acetate 22.5 Milligrams (mg)
Started | 107
Completed | 64
Not Completed | 43
Not completed — Adverse Event | 2
Not completed — Death | 9
Not completed — Lost to Follow-up | 1
Not completed — Progressive Disease | 22
Not completed — Protocol Violation | 2
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 5

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAF) :The SAF consisted of all participants who received at least 1 eligard injection and any follow-up safety information was available.
Arm/Group | Leuprolide Acetate 22.5 Milligrams (mg)
Number analyzed (Participants) | 106
Age, Continuous [Mean (Standard Deviation); unit: Years] | 72.2 (7.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 106
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 106
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 106
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Prostate-specific antigen (PSA) Level at Initial Diagnosis [Mean (Standard Deviation); unit: Nanogram per milliliter (ng/mL)] — Population: SAF population with available data.
  Nanogram per milliliter (ng/mL)
    number analyzed (Participants) | 103
    (all) | 315.05 (989.552)
EuroQol-5 Dimension-5 Level (EQ-5D-5L) Health State Utility Index Score (Japan) [Mean (Standard Deviation); unit: Score on a scale] — EQ-5D-5L is a standardized instrument for use as a measure of health outcome and provides a simple descriptive profile and a single index value for health status. EQ-5D-5L consists of 2 pages comprising the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension of the EQ-5D-5L has 5 levels and the participant was asked to indicate his health state by ticking the box with the most appropriate statement. Index scores were generated using Japan value sets. Scores ranged from -0.111 to 1. Higher scores indicate better health state. Population: Full analysis set (FAS): The FAS consisted of all participants who were enrolled and received at least 1 dose of ELIGARD and have at least 1 post baseline measurement of PSA and testosterone levels.
  Score on a scale
    number analyzed (Participants) | 105
    (all) | 0.8162 (0.18916)
EQ-5D-5L Index Score (UK) [Mean (Standard Deviation); unit: Score on a scale] — EQ-5D-5L is a standardized instrument for use as a measure of health outcome and provides a simple descriptive profile and a single index value for health status. EQ-5D-5L consists of 2 pages comprising the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension of the EQ-5D-5L has 5 levels and the participant was asked to indicate his health state by ticking the box with the most appropriate statement. Index scores were generated using UK value sets. Scores ranged from -0.594 to 1. Higher scores indicate better health state. Population: FAS population
  Score on a scale
    number analyzed (Participants) | 105
    (all) | 0.8040 (0.25853)
EQ-5D-5L Index Score (US) [Mean (Standard Deviation); unit: Score on a scale] — EQ-5D-5L is a standardized instrument for use as a measure of health outcome and provides a simple descriptive profile and a single index value for health status. EQ-5D-5L consists of 2 pages comprising the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension of the EQ-5D-5L has 5 levels and the participant was asked to indicate his health state by ticking the box with the most appropriate statement. Index scores were generated using US value sets. Scores ranged from -0.109 to 1. Higher scores indicate better health state. Population: FAS population
  Score on a scale
    number analyzed (Participants) | 105
    (all) | 0.8503 (0.18360)
EuroQol-5 Dimension-5 Level Health State Utility Index Visual Analogue Scale (EQ-5D02-EQ-VAS) [Mean (Standard Deviation); unit: Score on a scale] — The EQ5D02-EQ-VAS is a vertical VAS with values between 0 (worst imaginable health) and100 (best imaginable health), on which participants provide a global assessment of their health. Higher score indicate better health state. Population: FAS population
  Score on a scale
    number analyzed (Participants) | 105
    (all) | 78.8 (13.04)
European Organization for Research & Treatment of Cancer Quality of Life Questionnaire EORTCQLQ-PR25 [Mean (Standard Deviation); unit: Score on a scale] — EORTC QLQ-PR25 assesses urinary symptoms, bowel symptoms, treatment-related symptoms and sexual activity and functioning. It consist of 25 questions distributed on 6 domains: urinary symptoms (8 items), incontinence aid (1 item), bowel symptoms (4 items), hormonal treatment-related symptoms (HTRS) (6 items), sexual activity (2 items), and sexual functioning (4 items). Questions used 4 point scale (1 'Not at all' to 4 'Very much'). All raw domain scores are linearly transformed to a 0-100 scale, with higher scores reflecting either more symptoms or higher levels of activity or functioning. Population: FAS population with available data.
  Score on a scale
    Urinary Symptoms: number analyzed (Participants) | 102
    Urinary Symptoms | 29.38 (19.611)
    Incontinence Aid: number analyzed (Participants) | 55
    Incontinence Aid | 14.55 (26.265)
    Bowel Symptoms: number analyzed (Participants) | 105
    Bowel Symptoms | 7.06 (11.011)
    Hormonal Treatment Related Symptoms: number analyzed (Participants) | 105
    Hormonal Treatment Related Symptoms | 9.84 (11.690)
    Sexually Active: number analyzed (Participants) | 105
    Sexually Active | 13.02 (21.556)
    Sexual Function: number analyzed (Participants) | 51
    Sexual Function | 76.96 (7.447)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Eligard Related Adverse Events (AE)
Description: An AE was defined as any untoward medical occurrence in a participant administered a study drug or had undergone study procedures that did not necessarily have a causal relationship with this treatment. An AE was considered to be serious if, in the view of either the investigator or sponsor, it resulted in any of the following outcomes: resulted in death, was life-threatening, resulted in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions, resulted in congenital anomaly or birth defect, required inpatient hospitalization or led to prolongation of hospitalization, other medically important events. Drug-related AEs are AEs where causal relationships were at least a reasonable possibility as determined by the investigator.
Time Frame: From first dose of study drug up to 18 months
Population: SAF population
Measure: Number; unit: Participants
Groups:
- Leuprolide Acetate 22.5 mg: Participants received 22.5 mg of leuprolide acetate (eligard) by subcutaneous injection at baseline, month 3, 6, 9, 12 and 15.
Arm/Group | Leuprolide Acetate 22.5 mg
Number analyzed (Participants) | 106
Participants
  Drug-related adverse event | 15
  Drug-related serious adverse event | 2

2. Secondary Outcome: Percentage of Participants With Testosterone Levels Less Than (<) 20, 20-50 and Greater Than (>) 50 Nanogram Per Deciliter (ng/dL) at Month 12
Description: Testosterone level was summarized based on the percentage of participants with < 20 ng/dL, 20 to 50 ng/dL and > 50 ng/dL.
Time Frame: Month 12
Population: FAS population
Measure: Number; unit: Percentage of participants
Arm/Group | Leuprolide Acetate 22.5 mg
Number analyzed (Participants) | 105
Percentage of participants
  < 20 ng/dL | 51.4
  20 - 50 ng/dL | 12.4
  > 50 ng/dL | 1.9

3. Secondary Outcome: Percentage of Participants With Testosterone Levels < 20, 20-50 and > 50 ng/dL at Month 18
Description: as for outcome 2
Time Frame: Month 18
Population: FAS population
Measure: Number; unit: Percentage of participants
Arm/Group | Leuprolide Acetate 22.5 mg
Number analyzed (Participants) | 105
Percentage of participants
  < 20 ng/dL | 61.9
  20 - 50 ng/dL | 16.2
  > 50 ng/dL | 1.9

4. Secondary Outcome: Time to PSA Progression
Description: Time to PSA progression was defined as (date of ≥25 percentage (%) increase and ≥ 2 ng/mL absolute increase) - (date of first administration of ELIGARD 22.5 mg)/30, where PSA progression was defiined as 25% or greater increase and an absolute increase of 2 ng/mL, and confirmed by a second value at least 3 weeks later. Participants with more than 1 qualifying PSA progression were counted only once, and the earlier progression was accounted for time to progression analysis.
Time Frame: From first dose of study drug up to PSA progression (18 months)
Population: FAS population with available data.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Leuprolide Acetate 22.5 mg
Number analyzed (Participants) | 25
Months | 8.80 [6.10 to 9.20]

5. Secondary Outcome: Percentage of Participants With Greater Than or Equal to (≥) 30% PSA Percent Reduction From Baseline at Month 3, 6, 9, 12, 15, and 18
Description: PSA percent reduction (%) = ([PSA tested- baseline PSA]/baseline PSA)*100%. PSA level was summarized based on time to PSA progression and PSA percent reduction by ≥ 30% with respect to the level at baseline. Participants with more than 1 qualifying PSA progression were counted only once, and the earlier progression was accounted for time to progression analysis. PSA progression was defined as 25% or greater increase and an absolute increase of 2 nanogram per milliliter (ng/mL), and confirmed by a second value at least 3 weeks later.
Time Frame: Months 3, 6, 9, 12, 15 and 18
Population: FAS population with available data.
Measure: Number; unit: Percentage of participants
Arm/Group | Leuprolide Acetate 22.5 mg
Number analyzed (Participants) | 102
Percentage of participants
  Month 3 | 96.1
  Month 6: number analyzed (Participants) | 96
  Month 6 | 93.8
  Month 9: number analyzed (Participants) | 83
  Month 9 | 92.8
  Month 12: number analyzed (Participants) | 69
  Month 12 | 97.1
  Month 15: number analyzed (Participants) | 64
  Month 15 | 98.4
  Month 18: number analyzed (Participants) | 89
  Month 18 | 91.0

6. Secondary Outcome: Percentage of Participants With ≥50% PSA Percent Reduction From Baseline at Month 3, 6, 9, 12, 15, and 18
Description: PSA percent reduction (%) = ([PSA tested- baseline PSA]/baseline PSA)*100%. PSA level was summarized based on time to PSA progression and PSA percent reduction by ≥ 50% with respect to the level at baseline. Participants with more than 1 qualifying PSA progression were counted only once, and the earlier progression was accounted for time to progression analysis. PSA progression was defined as 25% or greater increase and an absolute increase of 2 ng/mL, and confirmed by a second value at least 3 weeks later.
Time Frame: Months 3, 6, 9, 12, 15 and 18
Population: FAS population with available data.
Measure: Number; unit: Percentage of participants
Arm/Group | Leuprolide Acetate 22.5 mg
Number analyzed (Participants) | 102
Percentage of participants
  Month 3 | 89.2
  Month 6: number analyzed (Participants) | 96
  Month 6 | 91.7
  Month 9: number analyzed (Participants) | 83
  Month 9 | 91.6
  Month 12: number analyzed (Participants) | 69
  Month 12 | 94.2
  Month 15: number analyzed (Participants) | 64
  Month 15 | 96.9
  Month 18: number analyzed (Participants) | 89
  Month 18 | 88.8

7. Secondary Outcome: Percentage of Participants With ≥90% PSA Percent Reduction From Baseline at Month 3, 6, 9, 12, 15, and 18
Description: PSA percent reduction (%) = ([PSA tested- baseline PSA]/baseline PSA)*100%. PSA level was summarized based on time to PSA progression and PSA percent reduction by ≥ 90%, with respect to the level at baseline. Participants with more than 1 qualifying PSA progression were counted only once, and the earlier progression was accounted for time to progression analysis. PSA progression was defined as 25% or greater increase and an absolute increase of 2 ng/mL, and confirmed by a second value at least 3 weeks later.
Time Frame: Months 3, 6, 9, 12, 15 and 18
Population: FAS population with available data.
Measure: Number; unit: Percentage of participants
Arm/Group | Leuprolide Acetate 22.5 mg
Number analyzed (Participants) | 102
Percentage of participants
  Month 3 | 69.6
  Month 6: number analyzed (Participants) | 96
  Month 6 | 77.1
  Month 9: number analyzed (Participants) | 83
  Month 9 | 77.1
  Month 12: number analyzed (Participants) | 69
  Month 12 | 81.2
  Month 15: number analyzed (Participants) | 64
  Month 15 | 79.7
  Month 18: number analyzed (Participants) | 89
  Month 18 | 68.5

8. Secondary Outcome: Change From Baseline in EQ-5D-5L Health State Utility Index Score (Japan) at Months 6, 12 and 18
Description: EQ-5D-5L is a standardized instrument for use as a measure of health outcome and provides a simple descriptive profile and a single index value for health status. EQ-5D-5L is designed for self-completion by respondents and consists of 2 pages comprising the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension of the EQ-5D-5L has 5 levels (no problems, slight problems, moderate problems, severe problems, and extreme problems) and the participant was asked to indicate his health state by ticking the box with the most appropriate statement. Index scores were generated using Japan value sets. Scores ranged from -0.111 to 1. Higher scores indicate better health state.
Time Frame: Baseline, months 6, 12 and 18
Population: FAS population with available data.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Leuprolide Acetate 22.5 mg
Number analyzed (Participants) | 95
Score on a scale
  Month 6 | -0.0047 (0.16874)
  Month 12: number analyzed (Participants) | 68
  Month 12 | -0.0093 (0.14456)
  Month 18: number analyzed (Participants) | 81
  Month 18 | -0.0262 (0.17520)

9. Secondary Outcome: Change From Baseline in EQ-5D-5L Health Status Utility Index Score (UK) at Months 6, 12 and 18
Description: EQ-5D-5L is a standardized instrument for use as a measure of health outcome and provides a simple descriptive profile and a single index value for health status. EQ-5D-5L is designed for self-completion by respondents and consists of 2 pages comprising the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension of the EQ-5D-5L has 5 levels (no problems, slight problems, moderate problems, severe problems, and extreme problems) and the participant was asked to indicate his health state by ticking the box with the most appropriate statement. Index scores were generated using UK value sets. Scores ranged from -0.594 to 1. Higher scores indicate better health state.
Time Frame: Baseline, months 6, 12 and 18
Population: FAS population with available data.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Leuprolide Acetate 22.5 mg
Number analyzed (Participants) | 95
Score on a scale
  Month 6 | 0.0055 (0.21662)
  Month 9: number analyzed (Participants) | 68
  Month 9 | -0.0051 (0.16493)
  Month 18: number analyzed (Participants) | 81
  Month 18 | -0.0259 (0.23831)

10. Secondary Outcome: Change From Baseline in EQ-5D-5L Health Status Utility Index Score (US) at Months 6, 12 and 18
Description: EQ-5D-5L is a standardized instrument for use as a measure of health outcome and provides a simple descriptive profile and a single index value for health status. EQ-5D-5L is designed for self-completion by respondents and consists of 2 pages comprising the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension of the EQ-5D-5L has 5 levels (no problems, slight problems, moderate problems, severe problems, and extreme problems) and the participants was asked to indicate his health state by ticking the box with the most appropriate statement. Index scores were generated using US value sets. Scores ranged from -0.109 to 1. Higher scores indicate better health state.
Time Frame: Baseline, months 6, 12 and 18
Population: FAS population with available data.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Leuprolide Acetate 22.5 mg
Number analyzed (Participants) | 95
Score on a scale
  Month 6 | 0.0017 (0.15819)
  Month 9: number analyzed (Participants) | 68
  Month 9 | -0.0047 (0.12477)
  Month 18: number analyzed (Participants) | 81
  Month 18 | -0.0191 (0.16934)

11. Secondary Outcome: Change From Baseline in EQ-5D02-EQ-VAS Score at Months 6, 12 and 18
Description: The EQ5D02-EQ-VAS is a vertical VAS with values between 0 (worst imaginable health) and 100 (best imaginable health), on which participants provide a global assessment of their health. Higher score indicate better health state.
Time Frame: Baseline, months 6, 12 and 18
Population: FAS population with available data.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Leuprolide Acetate 22.5 mg
Number analyzed (Participants) | 96
Score on a scale
  Month 6 | 1.3 (14.72)
  Month 9: number analyzed (Participants) | 69
  Month 9 | 2.1 (11.92)
  Month 18: number analyzed (Participants) | 82
  Month 18 | 2.0 (15.65)

12. Secondary Outcome: Change From Baseline in EORTC QLQ-PR25 Score at Months 6, 12 and 18
Description: EORTC QLQ-PR25 is a prostate cancer module for the assessment of health-related quality of life (HRQoL). EORTC QLQ-PR25 is designed for self-completion by respondents and assesses urinary symptoms, bowel symptoms, treatment-related symptoms and sexual activity and functioning. The rule of scoring for EORTC QLQ-PR25 follows instruction of EORTC QLQ-PR25 Scoring Manual 2.0. It consist of 25 questions distributed on 6 domains: urinary symptoms (8 items), incontinence aid (1 item), bowel symptoms (4 items), hormonal treatment-related symptoms (HTRS) (6 items), sexual activity (2 items), and sexual functioning (4 items). Questions used 4 point scale (1 'Not at all' to 4 'Very much'). All raw domain scores are linearly transformed to a 0-100 scale, with higher scores reflecting either more symptoms (urinary, bowel, hormonal treatment-related symptoms) or higher levels of activity or functioning (sexual).
Time Frame: Baseline, months 6, 12 and 18
Population: FAS population with available data.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Leuprolide Acetate 22.5 mg
Number analyzed (Participants) | 96
Score on a scale
  Week 6: Urinary Symptoms: number analyzed (Participants) | 94
  Week 6: Urinary Symptoms | -4.84 (15.669)
  Week 6: Incontinence Aid: number analyzed (Participants) | 32
  Week 6: Incontinence Aid | -5.21 (28.220)
  Week 6: Bowel Symptoms | -2.17 (8.311)
  Week 6: HTRS | 3.27 (11.008)
  Week 6: Sexually Active | -6.08 (17.290)
  Week 6: Sexual Function: number analyzed (Participants) | 26
  Week 6: Sexual Function | -1.44 (11.362)
  Week 12: Urinary Symptoms: number analyzed (Participants) | 66
  Week 12: Urinary Symptoms | -6.93 (15.237)
  Week 12: Incontinence Aid: number analyzed (Participants) | 18
  Week 12: Incontinence Aid | -11.11 (32.338)
  Week 12: Bowel Symptoms: number analyzed (Participants) | 69
  Week 12: Bowel Symptoms | -2.66 (9.533)
  Week 12: HTRS: number analyzed (Participants) | 69
  Week 12: HTRS | 2.14 (9.959)
  Week 12: Sexually Active: number analyzed (Participants) | 69
  Week 12: Sexually Active | -5.07 (16.983)
  Week 12: Sexual Function: number analyzed (Participants) | 23
  Week 12: Sexual Function | -2.99 (14.823)
  Week 18: Urinary Symptoms: number analyzed (Participants) | 78
  Week 18: Urinary Symptoms | -4.06 (15.370)
  Week 18: Incontinence Aid: number analyzed (Participants) | 20
  Week 18: Incontinence Aid | 1.67 (31.484)
  Week 18: Bowel Symptoms: number analyzed (Participants) | 80
  Week 18: Bowel Symptoms | 0.31 (9.036)
  Week 18: HTRS: number analyzed (Participants) | 81
  Week 18: HTRS | 4.68 (11.064)
  Week 18: Sexually Active: number analyzed (Participants) | 80
  Week 18: Sexually Active | -3.54 (23.334)
  Week 18: Sexual Function: number analyzed (Participants) | 22
  Week 18: Sexual Function | -8.52 (15.969)

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 18 months
Description: SAF Population
Arm/Group | Leuprolide Acetate 22.5 mg
All-Cause Mortality (participants affected / at risk) | 9/106
Serious Adverse Events (participants affected / at risk) | 31/106
Other Adverse Events (participants affected / at risk) | 42/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Leuprolide Acetate 22.5 mg (N=106)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Abdominal wall haematoma (Gastrointestinal disorders) | 1 (1)
Anal hypoaesthesia (Gastrointestinal disorders) | 1 (1)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Death (General disorders) | 3 (3)
Multiple organ dysfunction syndrome (General disorders) | 1 (1)
Peripheral swelling (General disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 4 (5)
Sepsis (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dementia (Nervous system disorders) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 2 (2)
Spinal cord compression (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Leuprolide Acetate 22.5 mg (N=106)
Anaemia (Blood and lymphatic system disorders) | 6 (6)
Upper respiratory tract infection (Infections and infestations) | 6 (8)
Prostatic specific antigen increased (Investigations) | 18 (18)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (14)
Hot flush (Vascular disorders) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2018-04-18): https://cdn.clinicaltrials.gov/large-docs/32/NCT03035032/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-28): https://cdn.clinicaltrials.gov/large-docs/32/NCT03035032/SAP_001.pdf